CLINICAL TRIAL: NCT02100696
Title: Phase III, Double-Blind, Placebo-Controlled, Multicenter Study of the Efficacy and Safety of Etrolizumab During Induction and Maintenance in Patients With Moderate to Severe Active Ulcerative Colitis Who Have Been Previously Exposed to TNF Inhibitors
Brief Title: A Study of the Efficacy and Safety of Etrolizumab in Participants With Ulcerative Colitis Who Have Been Previously Exposed to Tumor Necrosis Factor (TNF) Inhibitors
Acronym: HICKORY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA28950; 2013-004278-88 (EudraCT Number)
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase) (Experimental): Participants assigned to this arm will receive treatment with open-label etrolizumab 105 milligrams (mg) subcutaneous (SC) injection once every 4 weeks (Q4W) for 14 weeks during the induction phase.
  Interventions: Drug: Etrozulimab
- Cohort 2: Placebo (Double-Blind Induction Phase) (Placebo Comparator): Participants randomized to this arm will receive treatment with double-blind placebo SC injection Q4W for 14 weeks during the induction phase.
  Interventions: Drug: Placebo
- Cohort 2: Etrolizumab (Double-Blind Induction Phase) (Experimental): Participants randomized to this arm will receive treatment with double-blind etrolizumab 105 mg SC injection Q4W for 14 weeks during the induction phase.
  Interventions: Drug: Etrozulimab
- Placebo Responders: Placebo (Maintenance Phase) (Placebo Comparator): Participants who received placebo during the induction phase, Cohort 2: Placebo (Double-Blind Induction Phase), and achieve a clinical response with placebo at Week 14 will continue to receive blinded placebo from Week 16 up to Week 66 during the maintenance phase.
  Interventions: Drug: Placebo
- Etrolizumab Responders: Placebo (Maintenance Phase) (Placebo Comparator): Participants who received etrolizumab during the induction phase, Cohort 1: Etrolizumab (Open-Label Induction Phase) and Cohort 2: Etrolizumab (Double-Blind Induction Phase), and achieved a clinical response at Week 14 will be re-randomized by Week 16 for the double-blind maintenance phase. Clinical responders re-randomized to this arm will receive placebo SC injection Q4W from Week 16 up to Week 66.
  Interventions: Drug: Placebo
- Etrolizumab Responders: Etrolizumab (Maintenance Phase) (Experimental): Participants who received etrolizumab during the induction phase, Cohort 1: Etrolizumab (Open-Label Induction Phase) and Cohort 2: Etrolizumab (Double-Blind Induction Phase), and achieved a clinical response at Week 14 will be re-randomized by Week 16 for the double-blind maintenance phase. Clinical responders re-randomized to this arm will receive etrolizumab 105 mg SC injection Q4W from Week 16 up to Week 66.
  Interventions: Drug: Etrozulimab

INTERVENTIONS:
Drug: Etrozulimab — Participants will receive 105 mg etrolizumab administered by SC injection Q4W.
  Other Names: PRO145223; RO5490261; RG7413
  Arms: Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase); Cohort 2: Etrolizumab (Double-Blind Induction Phase); Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Drug: Placebo — Participants will receive placebo (matched with etrolizumab) administered by SC injection Q4W.
  Arms: Cohort 2: Placebo (Double-Blind Induction Phase); Etrolizumab Responders: Placebo (Maintenance Phase); Placebo Responders: Placebo (Maintenance Phase)

SUMMARY:
This Phase III, double-blind, placebo-controlled, multicenter study will investigate the efficacy and safety of etrolizumab during induction and maintenance of remission compared with placebo in the treatment of participants with moderately to severely active ulcerative colitis (UC) who have been previously exposed to TNF inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC established at least 3 months prior to Day 1
* Moderately to severely active UC as determined by the Mayo Clinic Score (MCS) assessment
* Treatment within 5 years prior to screening with one or two induction regimens that contain TNF inhibitors (including TNF inhibitor biosimilars)
* Washout of anti-TNF therapy for at least 8 weeks preceding Day 1
* Background regimen for UC may include oral 5-aminosalicylic acid (5-ASA), oral corticosteroids, budesonide, probiotics, azathioprine (AZA), 6-mercaptopurine (6-MP), or methotrexate (MTX) if doses have been stable during the screening period
* Use of highly effective contraception as defined by the protocol
* Must have received a colonoscopy within the past year or be willing to undergo a colonoscopy in lieu of a flexible sigmoidoscopy at screening

Exclusion Criteria:

* A history of or current conditions and diseases affecting the digestive tract, such as indeterminate colitis, suspicion of ischemic colitis, radiation colitis, or microscopic colitis, Crohn's disease, fistulas or abdominal abscesses, colonic mucosal dysplasia, intestinal obstruction, toxic megacolon, or unremoved adenomatous colonic polyps
* Prior or planned surgery for UC
* Past or present ileostomy or colostomy
* Any prior treatment with etrolizumab or other anti-integrin agents (including natalizumab, vedolizumab, and efalizumab)
* Any prior treatment with anti-adhesion molecules (e.g. anti-MAdCAM-1)
* Any prior treatment with rituximab
* Any treatment with tofacitinib during screening
* Congenital or acquired immune deficiency, chronic hepatitis B or C infection, human immunodeficiency virus (HIV) positive, or history of tuberculosis (active or latent)
* Evidence of or treatment for Clostridium difficile or clinically significant cytomegalovirus (CMV) colitis within 60 days prior to Day 1
* Evidence of or treatment for other intestinal pathogens within 30 days prior to Day 1
* History of recurrent opportunistic infections and/or severe disseminated viral infections
* History of organ transplant
* Any major episode of infection requiring treatment with intravenous (IV) antibiotics within 8 weeks prior to screening or oral antibiotics within 4 weeks prior to screening
* Received a live attenuated vaccine within 4 weeks prior to Day 1

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2014-05-21 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (184):
- United States (38):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Diego Medical Center, La Jolla, California
  - Clinical Applications Laboratories, Inc., San Diego, California
  - Precision Research Institute, LLC, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Rocky Mountain Gastroenterology Associates, Denver, Colorado
  - Rocky Mountain Gastroenterology Associates, P.L.L.C.; Gastroenterology, Lakewood, Colorado
  - FQL Research, LLC, Miramar, Florida
  - Center For Digestive Health, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Northwestern University Feinberg School Of Medicine, Chicago, Illinois
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Massachusetts General Hospital; Crohn's & Colitis Center, Boston, Massachusetts
  - University of Michigan; Michigan Institute for Clinical and Health Research (MICHR), Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Kansas City Research Institute, LLC, Kansas City, Missouri
  - Clinica Peruano Americana S.A., Great Neck, New York
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Consultants for Clinical Research Inc., Cincinnati, Ohio
  - UC Health, LLC., Cincinnati, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Gastroenterology Center of the Midsouth, P.C., Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Tyler Research Institute, LLC, Tyler, Texas
  - Ericksen Research and Development, Clinton, Utah
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Digestive and Liver Disease Specialists, Ltd., Norfolk, Virginia
  - McGuire Research Institute; Gastroenterology, Richmond, Virginia
  - Washington Gastroenterology, Bellevue, Washington
- Hospital Provincial del Centenario, Rosario, Argentina
- Australia (8):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Launceston General Hospital; Gastroenterology Research, Launceston, Tasmania
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Footscray Hospital; Gastroenterology, Footscray, Victoria
  - St Frances Xavier Cabrini Hospital, Malvern, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (3):
  - Klinikum Klagenfurt am Wörtersee; Acute geriatric care, Klagenfurt
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Belgium (8):
  - Imeldaziekenhuis, Bonheiden
  - CHU St Pierre (St Pierre), Brussels
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
  - AZ Sint Elisabeth Herentals, Herentals
  - UZ Leuven; Neurology, Leuven
  - CHU de Liège; Tour de Pathologie, Liège
  - AZ Delta (Stedelijk Ziekenhuis), Roeselare
- Brazil (9):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva Ltda, Goiânia, Goiás
  - Hospital Felicio Rocho, Belo Horizonte, Minas Gerais
  - Centro Digestivo de Curitiba, Curitiba, Paraná
  - Hospital Universitario Clementino Fraga Filho - UFRJ, Rio de Janeiro, Rio de Janeiro
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre X, Porto Alegre, Rio Grande do Sul
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu, São Paulo
  - CAEP - Centro Avancado de Estudos e Pesquisas Ltda., Campinas, São Paulo
  - Hospital Estadual Mario Covas, Santo André, São Paulo
- Canada (10):
  - University of Calgary; Heritage Medical Research Clinic, Calgary, Alberta
  - Zeidler Ledcor Centre - University of Alberta; Division of Gasroenterology, Edmonton, Alberta
  - Pacific Gastroenterology Associates, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre; Gastroenterology Research, Halifax, Nova Scotia
  - Taunton Health Centre, Oshawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Toronto Digestive Disease Associates, Vaughan, Ontario
  - Hotel Dieu de Levis, Lévis, Quebec
  - Hôpital Maisonneuve - Rosemont, Montreal, Quebec
- Czechia (6):
  - Fakultni nemocnice Brno; Interni kardiologicka klinika, Brno
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Pardubicka krajska nemocnice, a.s., Pardubice
  - ISCARE a.s., Prague
  - Nemocnice Na Bulovce, Prague
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad Labem, o.z., Ocni oddeleni, Ústí nad Labem
- Denmark (2):
  - Ålborg Universitets Hospital; Gastromedicinsk, Aalborg
  - Rigshospitalet; Medicinsk gastroenterologisk klinik, København Ø
- France (11):
  - CHU Amiens - Hopital Sud; Pharmacie - Secteur des Essais cliniques, Amiens Cedex01
  - Hôpital Beaujon, Clichy
  - Hopital Claude Huriez - CHU Lille, Lille
  - Hôpital Nord - CHU Marseille; Gastroenterology and Hepatology, Marseille
  - CHU Nice - Hopital de l'Archet 2, Nice
  - Hôpital Saint-Louis, Paris
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque - USN, Pessac
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
  - Höpital Hautepierre; Pediatrie1, Strasbourg
  - CHU de Toulouse - Hôpital Rangueil, Toulouse
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (14):
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - DRK Kliniken Berlin Westend, Berlin
  - Universitaetsklinikum Erlangen, Erlangen
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Universitätsklinikum Freiburg; Innere Medizin I; Hämatologie, Onkologie und Stammzelltransplantation, Freiburg im Breisgau
  - Universitaetsklinikum Halle (Saale), Halle
  - Hamburgisches Forschungsinstitut fuer CED, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Gastroenterologie Eppendorfer Baum, Hamburg
  - Medizinische Hochschule Hannover; Klinik für Gastroenterologie, Hepatologie und Endokrinologie, Hanover
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Klinikum Mannheim GmbH Universitätsklinikum, Mannheim
  - Universitaetsklinikum Muenster, Münster
  - Universitaetsklinikum Ulm, Ulm
- Anticancer Hospital of Thessaliniki " Theagenio", Thessaloniki, Greece
- Hungary (12):
  - Bekes Megyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaza, Békéscsaba
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Eszak-Kozep-budai Centrum, Uj Szent Janos Korhaz es Szakrendelo, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont; Fázis I-es Klinikai Farmakológiai Vizsgálóhely, Budapest
  - Debreceni Egyetem, Debrecen
  - Markhot Ferenc Oktato Korhaz es Rendelointezet, Eger
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz; II. Belgyogyaszat, Miskolc
  - Pecsi Tudomanyegyetem, Pécs
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Israel (5):
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital - Ein Kerem; Neurosurgery, Jerusalem
  - Rabin Medical Center-Beilinson Campus; Gaucher Clinic, Genetics Institute, Petach Tiqwa
  - Kaplan Medical Center, Rehovot
  - Assaf Harofeh, Rishon LeZiyyon
- Italy (11):
  - Azienda Ospedaliera S. Orsola-Malpighi, Bologna, Emilia-Romagna
  - A.O.U. Policlinico di Modena, Modena, Emilia-Romagna
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli (Presidio Ospedale Sacco), Milan, Lombardy
  - Ospedale di Circolo; Neuropsichiatria Infantile, Rho, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese (MI), Lombardy
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliera Di Padova, Padua, Veneto
- Lithuania (2):
  - Hospital of Lithuanian University of Health. Sciences Kaunas Clinics, Kaunas
  - Vilnius University Hospital Santariskiu Clinic Public Insti, Vilnius
- Centro Regiomontano de Estudios Clínicos Roma S.C., Monterrey, Nuevo León, Mexico
- Netherlands (4):
  - Amsterdam UMC, Locatie VUMC; Neurology, Amsterdam
  - Amsterdam UMC Location AMC, Amsterdam
  - Rijnstate; Internal Medicine Department, Arnhem
  - Radboudumc, NL -nijmegen
- Poland (10):
  - Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz
  - Nzoz All-Medicus, Katowice
  - Gabinet Lekarski, Bartosz Korczowski, Rzeszów
  - Niepubliczny Zaklad Opieki Zdrowotnej SONOMED, Szczecin
  - Centrum Zdrowia MDM, Warsaw
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw
  - Nzoz Vivamed, Warsaw
  - PlanetMed, Wroclaw
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
  - EuroMediCare Szpital Specjalistyczny z Przychodnią we Wrocławiu, Wroclaw
- SC Euroclinic Hospital SA, Bucharest, Romania
- South Korea (8):
  - Kyungpook National University Hospital; Opthalmology, Daegu
  - Korea University Ansan Hospital, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center., Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
- Spain (6):
  - Fundacion Hospital de Alcorcon; Servicio de Digestivo, Alcorcón, Madrid
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (3):
  - Inselspital-Universitaetsspital Bern; Institut fuer Spitalpharmazie, Bern
  - Cliniques Universitaires Saint-Luc; Nephrology, Bern
  - Crohn-Colitis Zentrum Bern - Gemeinschaftspraxis Balsiger, Seibold und Partner, Bern
- United Kingdom (10):
  - Addenbrooke's Hospital, Cambridge
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - The Royal London Hospital, London
  - University College London Hospital, London
  - St Thomas Hospital, London
  - King's College London, London
  - Fairfield General Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham University Hospitals; QMC Campus, Nottingham
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Peyrin-Biroulet L, Hart A, Bossuyt P, Long M, Allez M, Juillerat P, Armuzzi A, Loftus EV Jr, Ostad-Saffari E, Scalori A, Oh YS, Tole S, Chai A, Pulley J, Lacey S, Sandborn WJ; HICKORY Study Group. Etrolizumab as induction and maintenance therapy for ulcerative colitis in patients previously treated with tumour necrosis factor inhibitors (HICKORY): a phase 3, randomised, controlled trial. Lancet Gastroenterol Hepatol. 2022 Feb;7(2):128-140. doi: 10.1016/S2468-1253(21)00298-3. Epub 2021 Nov 17. PMID 34798039
- [Derived] Sandborn WJ, Vermeire S, Tyrrell H, Hassanali A, Lacey S, Tole S, Tatro AR; Etrolizumab Global Steering Committee. Etrolizumab for the Treatment of Ulcerative Colitis and Crohn's Disease: An Overview of the Phase 3 Clinical Program. Adv Ther. 2020 Jul;37(7):3417-3431. doi: 10.1007/s12325-020-01366-2. Epub 2020 May 22. PMID 32445184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 184 centers in 24 countries.
Pre-assignment Details: A total of 609 participants were enrolled into the Induction phase of this study and the entire study. A subset (259) of these participants moved into the Maintenance phase of this study.
Period: Induction Phase
Arm/Group | Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase) | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase) | Placebo Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Started | 130 | 95 | 384 | 0 | 0 | 0
Completed | 115 | 90 | 358 | 0 | 0 | 0
Not Completed | 15 | 5 | 26 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 2 | 13 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Multiple Reasons | 5 | 2 | 8 | 0 | 0 | 0
Period: Maintenance Phase
Arm/Group | Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase) | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase) | Placebo Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Started | 0 | 0 | 0 | 27 | 115 | 117
Completed | 0 | 0 | 0 | 26 | 106 | 112
Not Completed | 0 | 0 | 0 | 1 | 9 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 4 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Multiple Reasons | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: A total of 609 participants were enrolled into the Induction phase of this study and the entire study. A subset (259) of these participants moved into the Maintenance phase of this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase) | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase) | Placebo Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase) | Total
Number analyzed (Participants) | 130 | 95 | 384 | 27 | 115 | 117 | 868
Age, Continuous [Mean (Standard Deviation); unit: years] — Induction Phase Population: Participants in the Induction Phase of this study.
  years
    number analyzed (Participants) | 130 | 95 | 384 | 0 | 0 | 0 | 609
    (all) | 39.5 (13.5) | 38.8 (13.9) | 40.7 (13.3) |  |  |  | 40.1 (13.4)
Age, Continuous [Mean (Standard Deviation); unit: years] — Maintenance Phase Population: Participants in the Maintenance Phase of this study.
  years
    number analyzed (Participants) | 0 | 0 | 0 | 27 | 115 | 117 | 259
    (all) |  |  |  | 43.1 (13.8) | 42.0 (13.5) | 40.0 (12.9) | 41.2 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Induction Phase Population: Participants in the Induction Phase of this study.
  Participants
    number analyzed (Participants) | 130 | 95 | 384 | 0 | 0 | 0 | 609
    Female | 52 | 41 | 160 |  |  |  | 253
    Male | 78 | 54 | 224 |  |  |  | 356
Sex: Female, Male [Count of Participants; unit: Participants] — Maintenance Phase Population: Participants in the Maintenance Phase of this study.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 27 | 115 | 117 | 259
    Female |  |  |  | 9 | 43 | 57 | 109
    Male |  |  |  | 18 | 72 | 60 | 150
Race/Ethnicity, Customized [Number; unit: Participants] — Induction Phase Population: Participants in the Induction Phase of this study.
  Participants
    Hispanic or Latino: number analyzed (Participants) | 130 | 95 | 384 | 0 | 0 | 0 | 609
    Hispanic or Latino | 4 | 5 | 30 |  |  |  | 39
    Not Hispanic or Latino: number analyzed (Participants) | 130 | 95 | 384 | 0 | 0 | 0 | 609
    Not Hispanic or Latino | 118 | 76 | 321 |  |  |  | 515
    Not Reported or Unknown: number analyzed (Participants) | 130 | 95 | 384 | 0 | 0 | 0 | 609
    Not Reported or Unknown | 8 | 14 | 33 |  |  |  | 55
    American Indian or Alaska Native: number analyzed (Participants) | 130 | 95 | 384 | 0 | 0 | 0 | 609
    American Indian or Alaska Native | 0 | 1 | 0 |  |  |  | 1
    Asian: number analyzed (Participants) | 130 | 95 | 384 | 0 | 0 | 0 | 609
    Asian | 6 | 5 | 26 |  |  |  | 37
    Black or African American: number analyzed (Participants) | 130 | 95 | 384 | 0 | 0 | 0 | 609
    Black or African American | 3 | 1 | 6 |  |  |  | 10
    White: number analyzed (Participants) | 130 | 95 | 384 | 0 | 0 | 0 | 609
    White | 109 | 73 | 304 |  |  |  | 486
    Other: number analyzed (Participants) | 130 | 95 | 384 | 0 | 0 | 0 | 609
    Other | 12 | 15 | 48 |  |  |  | 75
Race/Ethnicity, Customized [Number; unit: Participants] — Maintenance Phase Population: Participants in the Maintenance Phase of this study.
  Participants
    Hispanic or Latino: number analyzed (Participants) | 0 | 0 | 0 | 27 | 115 | 117 | 259
    Hispanic or Latino |  |  |  | 1 | 8 | 9 | 18
    Not Hispanic or Latino: number analyzed (Participants) | 0 | 0 | 0 | 27 | 115 | 117 | 259
    Not Hispanic or Latino |  |  |  | 21 | 95 | 94 | 210
    Not Reported or Unknown: number analyzed (Participants) | 0 | 0 | 0 | 27 | 115 | 117 | 259
    Not Reported or Unknown |  |  |  | 5 | 12 | 14 | 31
    Asian: number analyzed (Participants) | 0 | 0 | 0 | 27 | 115 | 117 | 259
    Asian |  |  |  | 2 | 5 | 5 | 12
    Black or African American: number analyzed (Participants) | 0 | 0 | 0 | 27 | 115 | 117 | 259
    Black or African American |  |  |  | 0 | 1 | 3 | 4
    White: number analyzed (Participants) | 0 | 0 | 0 | 27 | 115 | 117 | 259
    White |  |  |  | 20 | 96 | 92 | 208
    Other: number analyzed (Participants) | 0 | 0 | 0 | 27 | 115 | 117 | 259
    Other |  |  |  | 5 | 13 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Induction Phase: Percentage of Participants With Remission at Week 14, as Determined by the Mayo Clinic Score (MCS)
Description: The Mayo Clinic Score (MCS) ranges from 0 to 12 and is a composite of 4 assessments (each rated from 0-3): stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores represent greater disease severity. Remission was defined as MCS less than or equal to (≤)2 with individual subscores ≤1 and a rectal bleeding subscore of 0.
Time Frame: Week 14
Population: The Modified Intent-to-Treat (mITT) population was defined as all participants randomised in Cohort 2 who received at least one dose of study drug, with participants grouped according to the treatment assigned at randomisation.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase)
Number analyzed (Participants) | 95 | 384
Percentage of Participants | 6.3 | 18.5
Statistical Analysis 1: Comparison: Cohort 2: Placebo (Double-Blind Induction Phase) vs Cohort 2: Etrolizumab (Double-Blind Induction Phase); Test type: Superiority; p = 0.0033, Cochran-Mantel-Haenszel; Adjusted difference in response rates = 12.2, 95% CI 2-sided [3.95 to 17.67]

2. Primary Outcome: Maintenance Phase: Percentage of Participants With Remission at Week 66 Among Participants Who Had Achieved a Clinical Response at Week 14, as Determined by the MCS
Description: The MCS ranges from 0 to 12 and is a composite of 4 assessments (each rated from 0-3): stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores represent greater disease severity. Remission was defined as MCS less than or equal to (≤)2 with individual subscores ≤1 and a rectal bleeding subscore of 0. Clinical Response is MCS with ≥3-point decrease and 30% reduction from baseline as well as ≥1-point decrease in rectal bleeding subscore or an absolute rectal bleeding score of 0 or 1.
Time Frame: Week 66
Population: The Modified Intent-to-Treat (mITT) population was defined as all participants randomised in the maintenance phase who received at least one dose of study drug, with participants grouped according to the treatment assigned at randomisation.
Measure: Number; unit: Percentage of Participants
Arm/Group | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 114 | 112
Percentage of Participants | 20.2 | 24.1
Statistical Analysis 1: Comparison: Etrolizumab Responders: Placebo (Maintenance Phase) vs Etrolizumab Responders: Etrolizumab (Maintenance Phase); Test type: Superiority; p = 0.4956, Cochran-Mantel-Haenszel; Treatment Difference = 3.8, 95% CI 2-sided [-7.13 to 14.56]

3. Secondary Outcome: Induction Phase: Percentage of Participants With Clinical Remission at Week 14, as Determined by the MCS
Description: The MCS ranges from 0 to 12 and is a composite of 4 assessments (each rated from 0-3): stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores represent greater disease severity. Clinical Remission is MCS ≤2 with individual subscores ≤1.
Time Frame: Week 14
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase)
Number analyzed (Participants) | 95 | 384
Percentage of Participants | 6.3 | 18.8
Statistical Analysis 1: Comparison: Cohort 2: Placebo (Double-Blind Induction Phase) vs Cohort 2: Etrolizumab (Double-Blind Induction Phase); Test type: Superiority; p = 0.0028, Cochran-Mantel-Haenszel — Nominal P-value reported (not adjusted for multiplicity); Adjusted Difference in Remission Rates = 12.5, 95% CI 2-sided [4.19 to 17.94]

4. Secondary Outcome: Induction Phase: Percentage of Participants With Clinical Response at Week 14, as Determined by the MCS
Description: as for outcome 2
Time Frame: Week 14
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase)
Number analyzed (Participants) | 95 | 384
Percentage of Participants | 31.6 | 45.8
Statistical Analysis 1: Comparison: Cohort 2: Placebo (Double-Blind Induction Phase) vs Cohort 2: Etrolizumab (Double-Blind Induction Phase); Test type: Superiority; p = 0.0241, Cochran-Mantel-Haenszel — Multiplicity P-value reported (adjusted for multiplicity); Adjusted Difference in Response Rates = 14.3, 95% CI 2-sided [3.21 to 24.14]

5. Secondary Outcome: Induction Phase: Percentage of Participants With Improvement From Baseline in Endoscopic Appearance of the Mucosa at Week 14, as Determined by the MCS Endoscopic Subscore
Description: The MCS ranges from 0 to 12 and is a composite of 4 assessments (each rated from 0-3): stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores represent greater disease severity. Improvement in endoscopic appearance of the mucosa is Endoscopy subscore ≤1.
Time Frame: Baseline and Week 14
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase)
Number analyzed (Participants) | 95 | 384
Percentage of Participants | 25.3 | 33.3
Statistical Analysis 1: Comparison: Cohort 2: Placebo (Double-Blind Induction Phase) vs Cohort 2: Etrolizumab (Double-Blind Induction Phase); Test type: Superiority; p = 0.1605, Cochran-Mantel-Haenszel — Multiplicity P-value reported (adjusted for multiplicity); Adjusted Difference in Response Rates = 8.1, 95% CI 2-sided [-2.54 to 17.22]

6. Secondary Outcome: Induction Phase: Percentage of Participants With Endoscopic Remission at Week 14, as Determined by the MCS Endoscopic Subscore
Description: The MCS ranges from 0 to 12 and is a composite of 4 assessments (each rated from 0-3): stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores represent greater disease severity. Endoscopic Remission is Endoscopy subscore = 0.
Time Frame: Week 14
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase)
Number analyzed (Participants) | 95 | 384
Percentage of Participants | 9.5 | 17.2
Statistical Analysis 1: Comparison: Cohort 2: Placebo (Double-Blind Induction Phase) vs Cohort 2: Etrolizumab (Double-Blind Induction Phase); Test type: Superiority; p = 0.3881, Cochran-Mantel-Haenszel — Multiplicity P-value reported (adjusted for multiplicity); Adjusted Difference in Remission Rates = 7.6, 95% CI 2-sided [-1.22 to 13.66]

7. Secondary Outcome: Induction Phase: Percentage of Participants With Histologic Remission at Week 14, as Determined by the Nancy Histological Index
Description: Nancy Histological Index (NHI) is a 5-level classification ranging from grade 0 (No histologically significant disease) to grade 4 (severely active disease). Histologic remission is defined as a Nancy Histological Index of 0 or 1.
Time Frame: Week 14
Population: The Modified Intent-to-Treat (mITT) population was defined as all participants randomised in Cohort 2 who received at least one dose of study drug, with participants grouped according to the treatment assigned at randomisation. Data presented below is only for participants included in the actual analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase)
Number analyzed (Participants) | 80 | 310
Percentage of Participants | 25.0 | 29.7
Statistical Analysis 1: Comparison: Cohort 2: Placebo (Double-Blind Induction Phase) vs Cohort 2: Etrolizumab (Double-Blind Induction Phase); Test type: Superiority; p = 0.5879, Cochran-Mantel-Haenszel — Multiplicity P-value reported (adjusted for multiplicity); Adjusted Difference in Remission Rates = 4.9, 95% CI 2-sided [-6.78 to 14.69]

8. Secondary Outcome: Induction Phase: Change From Baseline to Week 6 in MCS Rectal Bleed Subscore
Description: Rectal bleeding data were collected via the participant's diaries and each day a participant provided a score from 0 to 3 according to the following definitions: 0 = no blood in the stool; 1 = streaks of blood with stool less than half the time; 2 = obvious blood with stool most of the time; 3 = blood alone passed. The Mayo Clinic Score (MCS) rectal bleeding subscore was calculated as the worst value of three days of daily diary scores closest to anchor dates at baseline and post-baseline. The data was considered non-parametric and was reported using RANK analysis of covariance (ANCOVA). Participants were stratified by concomitant treatment with corticosteroids or immunosuppressants at randomization and disease activity measured during screening (MCS ≤9/MCS ≥10); the model adjusted for these stratification factors along with the baseline rectal bleeding (RB) subscore.
Time Frame: Baseline and Week 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase)
Number analyzed (Participants) | 94 | 383
Score on a Scale | -0.4 (0.8) | -0.7 (0.9)
Statistical Analysis 1: Comparison: Cohort 2: Placebo (Double-Blind Induction Phase) vs Cohort 2: Etrolizumab (Double-Blind Induction Phase); Test type: Superiority; p = 0.0351, ANCOVA — Multiplicity P-value reported (adjusted for multiplicity); Difference in Unadjusted Means = -0.2, 95% CI 2-sided [-0.5 to -0.0]

9. Secondary Outcome: Induction Phase: Change From Baseline to Week 6 in MCS Stool Frequency Subscore
Description: Stool frequency data were collected via the participant's diaries and each day a participant provided a score from 0 to 3 according to the following definitions: 0 = normal number of stools; 1 = 1 to 2 more stools than normal; 2 = 3 to 4 more stools than normal; 3 = 5 or more stools than normal. The Mayo Clinic Score (MCS) stool frequency subscore was calculated as the average of three days daily diary scores closest to anchor dates at baseline and post-baseline. The data was considered non-parametric and was reported using RANK analysis of covariance (ANCOVA). Participants were stratified by concomitant treatment with corticosteroids or immunosuppressants at randomization and disease activity measured during screening (MCS ≤9/MCS ≥10); the model adjusted for these stratification factors along with the baseline stool frequency (SF) subscore.
Time Frame: Baseline and Week 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase)
Number analyzed (Participants) | 94 | 383
Score on a Scale | -0.5 (0.9) | -0.6 (1.0)
Statistical Analysis 1: Comparison: Cohort 2: Placebo (Double-Blind Induction Phase) vs Cohort 2: Etrolizumab (Double-Blind Induction Phase); Test type: Superiority; p = 0.2698, ANCOVA — Multiplicity P-value reported (adjusted for multiplicity); Difference in Unadjusted Means = -0.2, 95% CI 2-sided [-0.4 to 0.1]

10. Secondary Outcome: Induction Phase: Change From Baseline to Week 14 in UC Bowel Movement Signs and Symptoms, as Assessed by the Ulcerative Colitis Patient-Reported Outcome Signs and Symptoms (UC-PRO/SS) Questionnaire
Description: The UC-PRO questionnaire is collected in the e-diary and completed by participants for at least 9-12 consecutive days prior to a study visit. The UC-PRO is being reported in three domains; two domains are key endpoints and reported as UC-PRO Signs and Symptoms (UC-PRO/SS). The bowel domain score ranges from 0-27, with a higher score indicating a worse disease state.
Time Frame: Baseline and Week 14
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase)
Number analyzed (Participants) | 80 | 272
Score on a Scale | -3.6 (0.6) | -5.2 (0.3)
Statistical Analysis 1: Comparison: Cohort 2: Placebo (Double-Blind Induction Phase) vs Cohort 2: Etrolizumab (Double-Blind Induction Phase); Test type: Superiority; p = 0.2698, Mixed Models Analysis — Multiplicity P-value reported (adjusted for multiplicity); Difference in Least Square Means = -1.6, 95% CI 2-sided [-2.9 to -0.3]

11. Secondary Outcome: Induction Phase: Change From Baseline to Week 14 in UC Functional Symptoms, as Assessed by the UC-PRO/SS Questionnaire
Description: The UC-PRO questionnaire is collected in the e-diary and completed by participants for at least 9-12 consecutive days prior to a study visit. The UC-PRO is being reported in three domains; two domains are key endpoints and reported as UC-PRO Signs and Symptoms (UC-PRO/SS). The functional (abdominal symptoms) domain score ranges from 0-12, with a higher score indicating a worse disease state.
Time Frame: Baseline and Week 14
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase)
Number analyzed (Participants) | 80 | 272
Score on a Scale | -1.1 (0.2) | -1.5 (0.1)
Statistical Analysis 1: Comparison: Cohort 2: Placebo (Double-Blind Induction Phase) vs Cohort 2: Etrolizumab (Double-Blind Induction Phase); Test type: Superiority; p = 0.3881, Mixed Models Analysis — Multiplicity P-value reported (adjusted for multiplicity); Difference in Least Square Means = -0.5, 95% CI 2-sided [-1.0 to 0.0]

12. Secondary Outcome: Induction Phase: Change From Baseline to Week 14 in Health-Related Quality of Life, as Assessed by the Overall Score of the Inflammatory Bowel Disease Questionnaire (IBDQ)
Description: The IBDQ score is a Total Score summed up from across all 32 questions on the questionnaire. The Total Score range is from 32 to 224 with higher scores representing a better quality of life.
Time Frame: Baseline and Week 14
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase)
Number analyzed (Participants) | 74 | 293
Scores on a Scale | 28.4 (4.12) | 37.4 (2.17)
Statistical Analysis 1: Comparison: Cohort 2: Placebo (Double-Blind Induction Phase) vs Cohort 2: Etrolizumab (Double-Blind Induction Phase); Test type: Superiority; p = 0.0445, ANCOVA — Nominal P-value reported (not adjusted for multiplicity); Difference in Adjusted Means = 9.1, 95% CI 2-sided [0.2 to 17.9]

13. Secondary Outcome: Maintenance Phase: Percentage of Participants With Clinical Remission at Week 66 Among Participants Who Had Achieved Clinical Remission at Week 14, as Determined by the MCS
Description: The MCS ranges from 0 to 12 and is a composite of 4 assessments (each rated from 0-3): stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores represent greater disease severity. Remission was defined as MCS less than or equal to (≤)2 with individual subscores ≤1 and a rectal bleeding subscore of 0. Clinical Remission is MCS ≤2 with individual subscores ≤1.
Time Frame: Week 66
Population: The Modified Intent-to-Treat (mITT) population was defined as all participants randomised in the maintenance phase who received at least one dose of study drug, with participants grouped according to the treatment assigned at randomisation. Data presented below is only for participants included in the actual analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 44 | 42
Percentage of Participants | 36.4 | 38.1
Statistical Analysis 1: Comparison: Etrolizumab Responders: Placebo (Maintenance Phase) vs Etrolizumab Responders: Etrolizumab (Maintenance Phase); Test type: Superiority; p = 0.9959, Cochran-Mantel-Haenszel — Nominal P-value reported (not adjusted for multiplicity); Adjusted Difference in Remission Rates = 0.1, 95% CI 2-sided [-19.67 to 19.88]

14. Secondary Outcome: Maintenance Phase: Percentage of Participants With Clinical Remission at Week 66, as Determined by the MCS
Description: as for outcome 13
Time Frame: Week 66
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 114 | 112
Percentage of Participants | 21.1 | 25.0
Statistical Analysis 1: Comparison: Etrolizumab Responders: Placebo (Maintenance Phase) vs Etrolizumab Responders: Etrolizumab (Maintenance Phase); Test type: Superiority; p = 0.5014, Cochran-Mantel-Haenszel — Nominal P-value reported (not adjusted for multiplicity); Adjusted Difference in Remission Rates = 3.8, 95% CI 2-sided [-7.26 to 14.70]

15. Secondary Outcome: Maintenance Phase: Percentage of Participants With Remission at Week 66 Among Participants Who Had Achieved Remission at Week 14, as Determined by the MCS
Description: The MCS ranges from 0 to 12 and is a composite of 4 assessments (each rated from 0-3): stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores represent greater disease severity. Remission was defined as MCS less than or equal to (≤)2 with individual subscores ≤1 and a rectal bleeding subscore of 0.
Time Frame: Week 66
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 44 | 41
Percentage of Participants | 34.1 | 36.6
Statistical Analysis 1: Comparison: Etrolizumab Responders: Placebo (Maintenance Phase) vs Etrolizumab Responders: Etrolizumab (Maintenance Phase); Test type: Superiority; p = 0.9538, Cochran-Mantel-Haenszel — Nominal P-value reported (not adjusted for multiplicity); Adjusted Difference in Remission Rates = 0.6, 95% CI 2-sided [-19.08 to 20.35]

16. Secondary Outcome: Maintenance Phase: Percentage of Participants With Improvement From Baseline in Endoscopic Appearance of the Mucosa at Week 66, as Determined by the MCS Endoscopic Subscore
Description: as for outcome 5
Time Frame: Baseline and Week 66
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 114 | 112
Percentage of Participants | 21.1 | 35.7
Statistical Analysis 1: Comparison: Etrolizumab Responders: Placebo (Maintenance Phase) vs Etrolizumab Responders: Etrolizumab (Maintenance Phase); Test type: Superiority; p = 0.0153, Cochran-Mantel-Haenszel — Nominal P-value reported (not adjusted for multiplicity); Adjusted Difference in Response Rates = 14.5, 95% CI 2-sided [2.66 to 25.78]

17. Secondary Outcome: Maintenance Phase: Percentage of Participants With Histologic Remission at Week 66, as Determined by the Nancy Histological Index
Description: as for outcome 7
Time Frame: Week 66
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 92 | 91
Percentage of Participants | 14.1 | 30.8
Statistical Analysis 1: Comparison: Etrolizumab Responders: Placebo (Maintenance Phase) vs Etrolizumab Responders: Etrolizumab (Maintenance Phase); Test type: Superiority; p = 0.0073, Cochran-Mantel-Haenszel — Nominal P-value reported (not adjusted for multiplicity); Adjusted Difference in Remission Rates = 16.8, 95% CI 2-sided [4.44 to 28.41]

18. Secondary Outcome: Maintenance Phase: Percentage of Participants With Endoscopic Remission at Week 66, as Determined by the MCS Endoscopic Subscore
Description: as for outcome 6
Time Frame: Week 66
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 114 | 112
Percentage of Participants | 11.4 | 23.2
Statistical Analysis 1: Comparison: Etrolizumab Responders: Placebo (Maintenance Phase) vs Etrolizumab Responders: Etrolizumab (Maintenance Phase); Test type: Superiority; p = 0.0174, Cochran-Mantel-Haenszel — Nominal P-value reported (not adjusted for multiplicity); Adjusted Difference in Remission Rates = 11.9, 95% CI 2-sided [1.87 to 21.71]

19. Secondary Outcome: Maintenance Phase: Percentage of Participants With Corticosteroid-Free Clinical Remission at Week 66 Among Participants Who Were Receiving Corticosteroids at Baseline, as Determined by the MCS
Description: The MCS ranges from 0 to 12 and is a composite of 4 assessments (each rated from 0-3): stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores represent greater disease severity. Corticosteroid-Free analysis was conducted only on a subgroup of participants who were randomized into the maintenance phase and receiving Corticosteroids (CS) at baseline. Participants were defined as being off CS if they had no record of taking CS on the date that was 24 weeks prior to Week 66.
Time Frame: Week 66
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 55 | 54
Percentage of Participants | 12.7 | 20.4
Statistical Analysis 1: Comparison: Etrolizumab Responders: Placebo (Maintenance Phase) vs Etrolizumab Responders: Etrolizumab (Maintenance Phase); Test type: Superiority; p = 0.3015, Cochran-Mantel-Haenszel — Nominal P-value reported (not adjusted for multiplicity); Adjusted Difference in Remission Rates = 7.3, 95% CI 2-sided [-6.83 to 21.60]

20. Secondary Outcome: Maintenance Phase: Percentage of Participants With Corticosteroid-Free Remission at Week 66 Among Participants Who Were Receiving Corticosteroids at Baseline, as Determined by the MCS
Description: as for outcome 19
Time Frame: Week 66
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 55 | 54
Percentage of Participants | 10.9 | 18.5
Statistical Analysis 1: Comparison: Etrolizumab Responders: Placebo (Maintenance Phase) vs Etrolizumab Responders: Etrolizumab (Maintenance Phase); Test type: Superiority; p = 0.2787, Cochran-Mantel-Haenszel — Nominal P-value reported (not adjusted for multiplicity); Adjusted Difference in Remission Rates = 7.4, 95% CI 2-sided [-6.23 to 21.17]

21. Secondary Outcome: Maintenance Phase: Change From Baseline to Week 66 in UC Bowel Movement Signs and Symptoms, as Assessed by the UC-PRO/SS Questionnaire
Description: as for outcome 10
Time Frame: Baseline and Week 66
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 83 | 83
Score on a Scale | -6.3 (0.6) | -7.8 (0.6)
Statistical Analysis 1: Comparison: Etrolizumab Responders: Placebo (Maintenance Phase) vs Etrolizumab Responders: Etrolizumab (Maintenance Phase); Test type: Superiority; p = 0.0763, Mixed Models Analysis — Nominal P-value reported (not adjusted for multiplicity); Difference in Least Square Means = -1.5, 95% CI 2-sided [-3.1 to 0.2]

22. Secondary Outcome: Maintenance Phase: Change From Baseline to Week 66 in UC Functional Symptoms, as Assessed by the UC-PRO/SS Questionnaire
Description: as for outcome 11
Time Frame: Baseline and Week 66
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 83 | 83
Score on a Scale | -1.8 (0.3) | -2.0 (0.3)
Statistical Analysis 1: Comparison: Etrolizumab Responders: Placebo (Maintenance Phase) vs Etrolizumab Responders: Etrolizumab (Maintenance Phase); Test type: Superiority; p = 0.5329, Mixed Models Analysis — Nominal P-value reported (not adjusted for multiplicity); Difference in Least Square Means = -0.2, 95% CI 2-sided [-1.0 to 0.5]

23. Secondary Outcome: Maintenance Phase: Change From Baseline to Week 66 in Health-Related Quality of Life, as Assessed by the Overall Score of the IBDQ
Description: The IBDQ is used to assess participant's health-related quality of life (QOL). The IBDQ score is a Total Score summed up from across all 32 questions on the questionnaire. The Total Score range is from 32 to 224 with higher scores representing a better quality of life.
Time Frame: Baseline and Week 66
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 99 | 99
Scores on a Scale | 57.2 (3.1) | 52.3 (3.1)
Statistical Analysis 1: Comparison: Etrolizumab Responders: Placebo (Maintenance Phase) vs Etrolizumab Responders: Etrolizumab (Maintenance Phase); Test type: Superiority; p = 0.2228, ANCOVA — Nominal P-value reported (not adjusted for multiplicity); Difference in Adjusted Means = -4.9, 95% CI 2-sided [-12.7 to 3.0]

24. Secondary Outcome: Number of Participants With at Least One Adverse Event by Severity, According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE v4.0)
Description: All Adverse Events (AEs) were graded for severity using the NCI-CTCAE v4.0. Any AE not specifically listed was assessed per the following 5 grades: Grade 1 = mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated. Grade 2 = moderate; minimal, local, or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living. Grade 3 = severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living. Grade 4 = life-threatening consequences or urgent intervention indicated. Grade 5 = death related to AE. Not all grades are appropriate for all AEs; some AEs have fewer than 5 options. The terms "severe" and "serious" are not synonymous and are independently assessed for each AE. Multiple occurrences of AEs were counted only once per participant at the highest (worst) grade.
Time Frame: From Baseline up to Week 78
Population: The Safety Population was defined as all participants who received at least one dose of study drug during the induction and maintenance phases. Participants were grouped by cohort and included in the treatment arm for the treatment most frequently received during the induction and maintenance phases.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase) | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase) | Placebo Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 130 | 95 | 384 | 27 | 114 | 112
Participants
  Grade 1 | 39 | 31 | 117 | 8 | 19 | 33
  Grade 2 | 38 | 26 | 97 | 14 | 64 | 45
  Grade 3 | 15 | 5 | 37 | 1 | 14 | 19
  Grade 4 | 0 | 1 | 2 | 0 | 0 | 1
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Adverse Events Leading to Study Drug Discontinuation
Time Frame: From Baseline up to Week 78
Population: as for outcome 24
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase) | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase) | Placebo Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 130 | 95 | 384 | 27 | 114 | 112
Participants | 2 | 1 | 12 | 4 | 9 | 10

26. Secondary Outcome: Number of Participants With Serious Infection-Related Adverse Events
Time Frame: From Baseline up to Week 78
Population: as for outcome 24
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase) | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase) | Placebo Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 130 | 95 | 384 | 27 | 114 | 112
Participants | 2 | 1 | 5 | 0 | 3 | 3

27. Secondary Outcome: Number of Participants With Infection-Related Adverse Events
Description: All Adverse Events (AEs) were graded for severity using the NCI-CTCAE v4.0. Any AE not specifically listed was assessed per the following 5 grades: Grade 1 = mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated. Grade 2 = moderate; minimal, local, or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living. Grade 3 = severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living. Grade 4 = life-threatening consequences or urgent intervention indicated. Not all grades are appropriate for all AEs; some AEs have fewer than 5 options. The terms "severe" and "serious" are not synonymous and are independently assessed for each AE. Multiple occurrences of AEs were counted only once per participant at the highest (worst) grade.
Time Frame: From Baseline up to Week 78
Population: as for outcome 24
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase) | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase) | Placebo Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 130 | 95 | 384 | 27 | 114 | 112
Participants | 38 | 29 | 100 | 13 | 44 | 58

28. Secondary Outcome: Number of Participants With Injection-Site Reaction-Related Adverse Events
Time Frame: From Baseline up to Week 78
Population: as for outcome 24
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase) | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase) | Placebo Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 130 | 95 | 384 | 27 | 114 | 112
Participants | 7 | 5 | 4 | 2 | 2 | 8

29. Secondary Outcome: Number of Participants With Hypersensitivity Reaction-Related Adverse Events
Time Frame: From Baseline up to Week 78
Population: as for outcome 24
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase) | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase) | Placebo Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 130 | 95 | 384 | 27 | 114 | 112
Participants | 0 | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Number of Participants With Malignancies
Time Frame: From Baseline up to Week 78
Population: as for outcome 24
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase) | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase) | Placebo Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 130 | 95 | 384 | 27 | 114 | 112
Participants | 0 | 0 | 2 | 0 | 0 | 2

31. Secondary Outcome: Number of Participants With Anti-Therapeutic Antibodies to Etrolizumab at Baseline and During the Study
Description: A tiered strategy was used to detect and characterize etrolizumab antibodies within this clinical study. When determining post baseline incidence, participants were considered to be ADA positive if they were ADA negative or had missing data at baseline but developed an ADA response following etrolizumab drug exposure (treatment-induced ADA response), or if they were ADA positive at baseline and the titer of one or more post baseline samples was at least 0.60 titer unit greater than the titer of the baseline sample (treatment-enhanced ADA response). Participants were considered to be ADA negative if they were ADA negative or had missing data at baseline and all post baseline samples were negative, or if they were ADA positive at baseline but did not have any post baseline samples with a titer that was at least 0.60 titer unit greater than the titer of the baseline sample (treatment unaffected).
Time Frame: Pre-dose at Baseline, Weeks 4, 14, 24, 44, and 66, and Early Termination/End of Safety Follow-Up (up to Week 78)
Population: Participants who received at least one dose of study treatment and had at least one baseline or post-baseline ATA result from at least one sample. For the Induction Phase, data for Cohorts 1 and 2 are combined to present the Etrolizumab Induction data for participants not randomised into the Maintenance phase.
Measure: Number; unit: Participants
Groups:
- Cohort 1: Etrolizumab (OLI Phase) + Cohort 2: Etrolizumab (Double-Blind Induction Phase): Cohort 1: Participants assigned to this arm will receive treatment with open-label etrolizumab 105 milligrams (mg) subcutaneous (SC) injection once every 4 weeks (Q4W) for 14 weeks during the induction phase.
  Cohort 2: Participants randomized to this arm will receive treatment with double-blind etrolizumab 105 mg SC injection Q4W for 14 weeks during the induction phase. Participants in this arm did not enter into the Maintenance phase of the study.
Arm/Group | Cohort 1: Etrolizumab (OLI Phase) + Cohort 2: Etrolizumab (Double-Blind Induction Phase) | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 286 | 114 | 112
Participants
  Baseline: number analyzed (Participants) | 286 | 114 | 110
  Baseline | 9 | 2 | 6
  Post-Baseline: number analyzed (Participants) | 284 | 114 | 112
  Post-Baseline | 68 | 35 | 28

32. Secondary Outcome: Etrolizumab Serum Trough Concentration (for Arms/Timepoints Above LLOQ)
Description: As per Protocol, the timepoints for each arm where more than a third of the samples were above the lower limit of quantification (LLOQ), full summary statistics (Mean and Standard Deviation) were reported. For timepoints below the LLOQ, only the Median and Max were reported as a separate outcome measure below.
Time Frame: Pre-dose (0 hour) at Baseline and Weeks 14, 24, 44 and 66
Population: All participants who received at least one dose of study drug and had evaluable PK data. For the Induction Phase, data for Cohorts 1 and 2 are combined to present the Etrolizumab Induction data for participants not randomised into the Maintenance phase.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (μg/mL)
Arm/Group | Cohort 1: Etrolizumab (OLI Phase) + Cohort 2: Etrolizumab (Double-Blind Induction Phase) | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
Number analyzed (Participants) | 251 | 113 | 110
micrograms per millilitre (μg/mL)
  Week 14 | 11.0 (4.66) | 12.7 (5.50) | 14.0 (6.12)
  Week 24: number analyzed (Participants) | 0 | 93 | 92
  Week 24 |  | 0.474 (0.742) | 9.55 (5.24)
  Week 44: number analyzed (Participants) | 0 | 0 | 71
  Week 44 |  |  | 10.7 (5.72)
  Week 66: number analyzed (Participants) | 0 | 0 | 59
  Week 66 |  |  | 16.2 (7.75)

33. Secondary Outcome: Etrolizumab Serum Trough Concentration (for Arms/Timepoints Below LLOQ)
Description: As per Protocol, the timepoints for each arm where more than a third of the samples were below the LLOQ only the Median and Max were reported.
Time Frame: Weeks 44 and 66
Population: All participants who received at least one dose of study drug and had evaluable PK data and were part of the timepoints that had more than a third of samples below LLOQ. For the Induction Phase, data for Cohorts 1 and 2 are combined to present the Etrolizumab Induction data for participants not randomised into the Maintenance phase.
Measure: Median (Full Range); unit: micrograms per millilitre (μg/mL)
Arm/Group | Etrolizumab Responders: Placebo (Maintenance Phase)
Number analyzed (Participants) | 113
micrograms per millilitre (μg/mL)
  Week 44: number analyzed (Participants) | 54
  Week 44 | 0.0400 [NA to 2.73] — As per Protocol, only the Median and Max were reported for timepoints where more than a third of the samples were below the LLOQ.
  Week 66: number analyzed (Participants) | 40
  Week 66 | 0.0400 [NA to 0.0400] — As per Protocol, only the Median and Max were reported for timepoints where more than a third of the samples were below the LLOQ.

ADVERSE EVENTS:
Time Frame: Baseline up until a maximum of 78 weeks.
Arm/Group | Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase) | Cohort 2: Placebo (Double-Blind Induction Phase) | Cohort 2: Etrolizumab (Double-Blind Induction Phase) | Placebo Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Placebo (Maintenance Phase) | Etrolizumab Responders: Etrolizumab (Maintenance Phase)
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/95 | 0/384 | 0/27 | 0/114 | 0/112
Serious Adverse Events (participants affected / at risk) | 11/130 | 5/95 | 20/384 | 2/27 | 7/114 | 11/112
Other Adverse Events (participants affected / at risk) | 38/130 | 31/95 | 115/384 | 20/27 | 78/114 | 78/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase) (N=130) | Cohort 2: Placebo (Double-Blind Induction Phase) (N=95) | Cohort 2: Etrolizumab (Double-Blind Induction Phase) (N=384) | Placebo Responders: Placebo (Maintenance Phase) (N=27) | Etrolizumab Responders: Placebo (Maintenance Phase) (N=114) | Etrolizumab Responders: Etrolizumab (Maintenance Phase) (N=112)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 6 (6) | 2 (3) | 10 (10) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pouchitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Uteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affect liability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Etrolizumab (Open-Label Induction (OLI) Phase) (N=130) | Cohort 2: Placebo (Double-Blind Induction Phase) (N=95) | Cohort 2: Etrolizumab (Double-Blind Induction Phase) (N=384) | Placebo Responders: Placebo (Maintenance Phase) (N=27) | Etrolizumab Responders: Placebo (Maintenance Phase) (N=114) | Etrolizumab Responders: Etrolizumab (Maintenance Phase) (N=112)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 10 (11)
Colitis ulcerative (Gastrointestinal disorders) | 9 (9) | 10 (10) | 36 (37) | 11 (11) | 46 (52) | 31 (32)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 6 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (7) | 7 (7)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 5 (6)
Fatigue (General disorders) | 8 (11) | 1 (1) | 10 (13) | 1 (1) | 4 (4) | 12 (13)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 5 (9)
Pyrexia (General disorders) | 5 (7) | 6 (8) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (9) | 5 (5)
Nasopharyngitis (Infections and infestations) | 12 (12) | 7 (8) | 33 (35) | 4 (5) | 17 (22) | 23 (33)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 5 (8) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 7 (7) | 33 (38) | 4 (6) | 8 (11) | 19 (26)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 10 (11) | 6 (8) | 22 (26) | 3 (3) | 10 (12) | 10 (10)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 8 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT02100696/Prot_002.pdf
  • Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT02100696/SAP_001.pdf